# Comprehensive analysis of the program: Salud Escolar

Unique Protocol ID: P86-19

4<sup>th</sup> August 2020



### COMPREHENSIVE ANALYSIS OF THE SALUD ESCOLAR PROGRAM IN MEXICO IMPACT ANALYSIS

#### Written informed consent letter for parents

Dear father / mother:

Your son/daughter has been selected to participate in the comprehensive evaluation study of the Salud Escolar: Escuelas Sanas y Activas. This document explains all aspects of the <u>impact analysis</u> component of this research study including purpose, procedures, the risks of the procedures, and the potential benefits. Once you have a clear idea about these components, you will be asked if you want your son / daughter to participate, if so, you will be asked to sign this authorization. After obtaining your authorization, we will also ask your son / daughter if he or she agrees to participate, if so, you will also be asked to sign an authorization.

ONCE READ, APPROVED AND SIGNED, PLEASE KEEP THE STUDY INFORMATION FOUND ON PAGES 1, 2 AND 3 AND SEND ONLY THE REMOVABLE SHEET (page 4) WITH YOUR DAUGHTER / SON TO SCHOOL.

**Purpose of the study:** The purpose of this study is to evaluate the effectiveness of the Salud Escolar: Escuelas Sanas y Activas program in promoting correct nutrition, adequate hydration, and physical activity in the school population of Mexico City.

**Study Procedures**: If you and your son / daughter decide to participate, we ask that you participate in the following activities:

- You will answer a questionnaire about sociodemographic characteristics of the home, food consumption habits and physical activity in your family that will take approximately 20 minutes. This questionnaire will be sent with your son / daughter for you to answer at home.
- Your son / daughter will answer a questionnaire about food (24- hour reminder) at school with an approximate duration of 30 minutes. This reminder will be applied twice, once at the start of the study, and the second time after 10 months.
- Trained and properly identified personnel will record the weight and height of your son / daughter at school, at the beginning of the study and after 10 months. Your son / daughter will fill out a beverage consumption diary for 3 days, at the start of the study and after 10 months.



-Your son / daughter will receive a portable motion recorder (accelerometer) that will be placed at hip height on the right side (Figure 1). This is a device that objectively measures the amount of movement your child performs during the day. The device will only record the general movement performed, it will not record where the child is, nor the type of activity he is doing. Using this meter does not alter your child's daily and / or academic activities. Monitoring with this device will last twenty-four hours (24 hours) for seven (7) consecutive days. Its use will be monitored daily at school and during the weekend and daily reminds to wear it will be sent via SMS or phone call. This measurement will be done at the start of the study and again 10 months later. The image on the right illustrates how your son / daughter should wear the accelerometer during the measurement period



Figure 1. Correct position of the movement meter on the right hip.

**Study risks**: The risk of this study is minimal for you or your son / daughter.

**Study Benefits**: You and your son / daughter will not receive any financial or other benefits for their participation. The information that you and your son / daughter provide us will be used to make recommendations to improve this Program.



Privacy Notice simplified: the main researcher of this study, Dra. Alejandra Jauregui de la Mota, is responsible for the treatment and protection of the personal data that you provide us, which will be protected in accordance with the provisions of the General Data Protection Law Personal in Possession of Obligatory Subjects. The personal data that we will request will be used exclusively for the purposes set forth in this document. You can request the correction of your data or that your data be removed from our databases or withdraw your consent for its use. In any of these cases we ask you to contact the researcher responsible for the project at the following email address: alejandra.jauregui@insp.mx

**Confidentiality**: All the information collected will be used for research purposes. All personal information about you or your family collected in this study will be strictly confidential. Your son / daughter's name will not be used in any type of publication. In all study files your son / daughter will be identified with a number and the name will be known only to the researcher. Neither your name nor that of your son / daughter will be used in scientific publications.

**Participation is voluntary**: Participation in the study is completely voluntary. If you or your son / daughter do not want to participate or want to withdraw after starting the study, this will not affect your and your child's relationship with researchers and educational institutions now or in the future.

**Contact Numbers:** If you have any questions, comments, or concerns regarding the project, please contact 10:00 a.m. to 5:00 p.m. in Mexico City, Mexico with Dr. Alejandra Jauregui de la Mota, researcher responsible for the project at the National Institute of Public Health, at the following telephone number (777) 329-30-00 extension 2373 or email: alejandra.jauregui@insp.mx

If you have general questions about your rights as a participant in a research study, you can contact the President of the Ethics and Research Committee of the National Institute of Public Health, Dr. Angélica Ángeles Llerenas, at: (777) 329-30-00 extension 7424 from Monday to Friday from 8:30 a.m. to 4:30 p.m. (Mexico time) or if you prefer you can write to the following email address: etica@correo.insp.mx



#### **REMOVABLE SHEET**

(You should only send this sheet with your daughter / son to school)

## INFORMED PARENT CONSENT AUTHORIZATION TO PARTICIPATE IN THE PROJECT "INTEGRAL ANALYSIS OF THE SALUD ESCOLAR PROGRAM IN MEXICO"

**Consent:** My son / daughter and I have discussed this with a member of the research team to my satisfaction. My son / daughter and I understand that our participation is voluntary. I have read this document and allow my son / daughter to enter this research study. Signing this document does not deprive me of my legal rights. I will receive a copy of this document.

| Student's name and surname: _ | | |
|-------------------------------|-----------------|------|
| Name of mother / father: | | |
| Telephone: | _ Home address: | |
| Mother's occupation: | | |
| School: | | |
| Signature | | |
| Mother / Father | | Date |

Institutional stamp
Approved Version: October 30, 2019
CI: 1633. Identifier Folio: S53
Copy stamped in file